CLINICAL TRIAL: NCT07069829
Title: Real-world, International, Multicentre, Non-interventional, Prospective Cohort to Assess Clinical and Patient-reported Outcomes in Adults With Moderate to Severe COPD Treated With Breztri/Trixeo in Routine Care Settings
Brief Title: Study of Clinical and Patient-reported Outcomes in Adults With Moderate to Severe COPD Treated With Breztri/Trixeo
Acronym: iCHOROS
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00128
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Moderate to Severe Chronic Obstructive Pulmonary Disease; Severe Exacerbations; BGF - Budesonide/Glycopyrrolate/Formoterol Fumarate
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic Obstructive Pulmonary Disease is a leading cause of global morbidity and mortality, especially in low- and middle-income countries. Exacerbations accelerate disease progression and increase the risk of death. Recent recommendations from the GOLD report emphasize the diagnosis of COPD and treatment planning based on a combination of lung function metrics, exacerbation history, and patient-reported symptoms. It is recommending the use of triple combination therapy (ICS+LABA+LAMA) such as BREZTRI/TRIXEO as one of the options in Group E patients. While BGF has demonstrated efficacy in controlled clinical trials, real-world evidence is needed to assess its impact on daily patient outcomes and quality of life.

The iCHOROS study is a real-world, international, multicenter, observational study aiming to evaluate changes in clinical and patient-reported outcomes in adults with moderate to severe COPD treated with BGF for 12 months in routine care settings across Latin America, Asia, and the Middle East & Africa. The study will provide valuable insights into the effectiveness and patient experience of BGF therapy in diverse, real-world populations

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease poses a major health challenge globally and is currently the third leading cause of death worldwide, resulting in approximately 3.23 million deaths annually. The impact of COPD is particularly pronounced in low- and middle-income countries where healthcare resources may be limited. COPD is characterized by a progressive decline in lung function, frequent exacerbations, and high morbidity and mortality rates. Exacerbations, which are acute worsening events of respiratory symptoms, play a critical role in disease progression. Hospitalized severe exacerbations markedly increase the risk of further exacerbations, a rapid decline in health status, and high short-term mortality rates. Roughly 20% of patients at GOLD stage 2 experience frequent exacerbations necessitating additional interventions, with risk increasing in GOLD stages 3 and 4.

Recent clinical guidelines from the Global Initiative for Chronic Obstructive Lung Disease (GOLD) emphasize a multidimensional assessment, incorporating lung function, prior exacerbation history, and patient-reported symptoms to guide treatment. The overall goal of COPD pharmacologic therapy is to reduce symptoms (including dyspnea), prevent exacerbations, improve exercise tolerance, and enhance quality of life. Triple inhaled therapy, consisting of an inhaled corticosteroid (ICS), long-acting muscarinic antagonist (LAMA), and long-acting β2-agonist (LABA), is recommended for patients in GOLD Group E who continue to experience exacerbations despite dual therapy. This approach has demonstrated beneficial effect in reducing mortality among high-risk, symptomatic COPD patients.

Breztri/Trixeo (BGF) is a fixed-dose triple combination of budesonide (ICS), glycopyrrolate (LAMA), and formoterol fumarate (LABA), administered via a metered dose inhaler utilizing Aerosphere™ delivery technology. BGF received regulatory approval from the FDA in July 2020 and the EMA in December 2020, based on phase III randomized controlled trials (RCTs) that established its efficacy in improving lung function and reducing moderate/severe exacerbations. These trials primarily measured lung function and exacerbation rates and also included secondary endpoints evaluating patient-reported outcomes (PROs). Despite these findings, there is a need for real-world evidence (RWE) to better understand the effectiveness, safety, and patient experience of BGF outside the controlled environment of RCTs.

The importance of capturing PROs-such as the COPD Assessment Test (CAT) and modified Medical Research Council (m-MRC) dyspnea scale-in both clinical trials and real-world studies is increasingly recognized in the literature and reflected in current GOLD recommendations. Observational, patient-centric studies in routine clinical practice can provide complementary insights to RCTs, particularly through direct and timely collection of PRO data. Such studies elucidate the real-life impact of COPD and its management on daily patient functioning and quality of life and are valuable to healthcare payers, practitioners, and patients themselves.

To address gaps in population diversity of earlier RCTs and to better understand the use of BGF in routine medical practice, the iCHOROS study is a non-interventional, prospective, multinational, multicenter observational cohort study designed to document clinical and patient-reported outcomes in COPD patients initiated on BGF. The study includes patients from diverse and often underrepresented regions, such as Latin America (Mexico, Argentina, Colombia, Central America and Caribbean, Costa Rica, Panama), Asia (Taiwan, Philippines, India, Vietnam, Malaysia, Indonesia, Thailand), and the Middle East and Africa (KSA, Kuwait, UAE, Egypt, Jordan). This design supports the collection of more generalizable and globally relevant data.

The primary objective of this study is to estimate the change in COPD health status using the mean change from baseline in CAT score after 12 weeks of BGF treatment. Secondary objectives include evaluating CAT score changes at weeks 26 and 52, determining the proportion of CAT responders at week 12, comparing moderate and severe exacerbation rates before and after BGF initiation, and describing patient satisfaction with inhaler devices across all visits. Additional endpoints include global impression of change and severity (PGI-C, PGI-S), BGF treatment patterns and reasons for discontinuation, changes in m-MRC score and spirometry parameters (FEV1, FVC, FEV1/FVC), as well as exploratory assessments of baseline clinical characteristics and cardiovascular events.

In accordance with real-world clinical practice, patient follow-up visits will occur at baseline, week 12, week 26, and week 52, with all treatments and diagnostic evaluations determined solely by the attending physician and local guidelines. Patients' demographics, vital signs, medical and exacerbation history, and medication use will be recorded at baseline. The decision to initiate BGF and all management is entirely at the physician's discretion, separate from study participation or informed consent. Study participation will cease upon discontinuation of BGF. The data collection is hybrid, using existing medical records and primary data from scheduled visits without altering the standard of care or providing investigational medication. The total duration for each patient is 52 weeks or until discontinuation of BGF, and the overall study timeframe is estimated at 21 months, including interim analyses for CAT score and exacerbation rate results as more than half the population reaches key visits. Overall, the iCHOROS study aims to comprehensively characterize real-world clinical and patient-reported outcomes associated with BGF, thus supporting better clinical decisions and patient-centered care for COPD worldwide.

ELIGIBILITY:
Inclusion Criteria:

The study will include patients who were prescribed BGF, but not yet initiated, according to the label (SmPC) and local market reimbursement criteria. Patients will only be included in the study if they meet the following inclusion criteria:

1. Patients diagnosed with COPD, at least 12 months before baseline, as assessed per physician's routine practice or as documented in the patient's chart.
2. Male or female patients aged over 30 years and under 80 years at the time of enrolment.
3. Patients providing a written Informed Consent* prior to inclusion to the study.

   *Prescription of BGF should be prior to the signed informed consent and the decision to prescribe this therapy is clearly separated from the physician's decision to include the patient in the current study.
4. Patients able and willing to read and to comprehend written instructions, and to comprehend and complete the questionnaires required by the protocol.

Exclusion Criteria:

Patients who meet any of the following criteria will not be eligible to participate in the study:

1. Patients with COPD due to documented α-1 antitrypsin deficiency.
2. Patients with recent (≤3 months) major cardiac or pulmonary events that required hospitalization (e.g., myocardial infarction, pulmonary embolism).
3. Patients previously treated with triple fixed-dose combination therapies 12 months before the screening visit or treated with Multiple Inhaled Triple Therapy (MITT) within the last 3 months before the screening visit.
4. Patients hospitalized due to COPD exacerbations within the last 30 days prior to enrolment.
5. Currently pregnant (or intending to become pregnant), breastfeeding, or lactating women.
6. Patients with a current diagnosis of asthma, active tuberculosis, lung cancer or lung metastasis, significant bronchiectasis, sarcoidosis, pulmonary fibrosis, pulmonary hypertension, interstitial lung diseases, or other active clinically significant pulmonary diseases.
7. Patients currently participating in a non-interventional observational trial that might, in the investigator's opinion, influence the assessment for the current study or participation in any interventional trial in the last 30 days prior to enrolment.
8. Patients with respiratory tract infection (including COVID-19 infection) ) that has not resolved ≤30 days prior to BGF MDI initiation and those exhibiting persistent long-COVID symptoms are excluded from the study.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study plans to enroll approximately 1,400 patients, accounting for an expected dropout rate or missing data of ~20%, to ensure that at least 1,120 patients complete the study.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
change from baseline in the COPD Assessment Test | 12 weeks
  Mean change from baseline in the COPD Assessment Test (CAT) scores after 12 weeks from treatment initiation

SECONDARY OUTCOMES:
CAT scores | 26 Weeks
  Mean change from baseline in CAT scores after 26 weeks of treatment
CAT scores | 52 weeks
  Mean change from baseline in CAT scores after 52 weeks of treatment
CAT scores | 12 weeks
  Percent of responders of the CAT achieving MCID ≥ 2 after 12 weeks of treatment compared to baseline.
TSQM - 9 Score | Baseline
  IQVIA Treatment Satisfaction Questionnaire for Medication-9 (TSQM-9)© scores at baseline
TSQM - 9 Score | 12 weeks
  IQVIA Treatment Satisfaction Questionnaire for Medication-9 (TSQM-9)© scores at 12 weeks
TSQM - 9 Score | 26 Weeks
  IQVIA Treatment Satisfaction Questionnaire for Medication-9 (TSQM-9)© scores at 26 weeks
TSQM - 9 Score | 52 weeks
  IQVIA Treatment Satisfaction Questionnaire for Medication-9 (TSQM-9)© scores at 52 weeks.
PGI-C Scale | 52 weeks
  Mean change from baseline in patient global impression of change (PGI-C) after 52 weeks from treatment initiation
PGI-S Scale | 12 weeks
  Mean change from baseline in COPD symptoms severity using the patient global impression of severity (PGI-S) after 12 weeks from treatment initiation
PGI-S Scale | 26 Weeks
  Mean change from baseline in COPD symptoms severity using the patient global impression of severity (PGI-S) after 26 weeks from treatment initiation
PGI-S Scale | 52 Weeks
  Mean change from baseline in COPD symptoms severity using the patient global impression of severity (PGI-S) after 52 weeks from treatment initiation
mMRC dyspnoea score | 12 weeks
  Mean change from baseline in mMRC dyspnoea score after 12 weeks from treatment initiation.
mMRC dyspnoea score | 26 Weeks
  Mean change from baseline in mMRC dyspnoea score (Appendix 6) after 26 weeks from treatment initiation.
mMRC dyspnoea score | 52 weeks
  Mean change from baseline in mMRC dyspnoea score (Appendix 6) after 52 weeks from treatment initiation.

CONTACTS AND LOCATIONS:
Locations (8):
- Saudi Arabia (2):
  - Research Site, Abhā
  - Research Site, Riyadh
- Taiwan (4):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Yunlin
- Vietnam (2):
  - Research Site, Hà Nội, Vietnam
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home